CLINICAL TRIAL: NCT05768321
Title: A Phase 1 Open-Label Study to Assess the Safety, Pharmacokinetics, and Preliminary Efficacy of GEC255 Oral Tablets in Subjects With Advanced Solid Tumors With KRAS p.G12C Mutation
Brief Title: Study of GEC255 in Subjects With Advanced Solid Tumors With KRAS p.G12C Mutation
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: GenEros Biopharma Hangzhou Ltd (Industry)
Responsible Party: Sponsor
Organization: GenEros Biopharma Ltd (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEC255-P1-01
Record Dates: First submitted 2023-02-15; First posted 2023-03-14 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GEC255 treatment (Experimental): Oral tablet(s), once daily in 28-day cycles
  Interventions: Drug: GEC255 tablets

INTERVENTIONS:
Drug: GEC255 tablets — Part 1: Dose escalation After initial starting dose cohort, daily dosages in subsequent cohorts are determined by cohort review committee.
  Part 2: Dose expansion Daily oral dosage RP2D based on data from Part 1

SUMMARY:
The overall objective of this Phase 1 study is to evaluate the safety, Pharmacokinetics (PK), and anti-tumor activity of daily oral dosing with GEC255 tablets in subjects with advanced solid tumor with Kirsten Rat Sarcoma (KRAS) p.G12C mutation. To determine the recommended Phase 2 dose (RP2D) based on assessments of multiple dose escalation and expansion in target cohorts.

DETAILED DESCRIPTION:
This First-in-human dose escalation and expansion study of GEC255 tablets in patients with advanced solid tumors with KRAS p.G12C mutation aims to evaluate the safety, tolerability, PK and preliminary efficacy of orally administered GEC255, to determine the MTD, DLT (if exists) and RP2D, and explore the potential biomarker associated with efficacy or drug resistance.

ELIGIBILITY:
Inclusion Criteria:

1. Has histologically or cytologically confirmed advance tumors with KRAS p.G12C mutation and has poor response to standard of care therapy or intolerant to standard of care therapies (chemotherapy, targeting therapy or immunotherapy).
2. As assessed by the investigator, the subject must have at least one measurable lesion that meets the definition of Response Evaluation Criteria in Solid Tumours (RECIST) 1.1 (subjects with only non-target lesions are allowed to be included in the dose escalation phase)
3. For the second part, subjects with non-small cell lung cancer must have received at least first-line platinum-based chemotherapy and/or immunotherapy /or anti-vascular therapy; subjects with colorectal cancer must have previously received second-line or above therapies and have tumor progression or recurrence. Except for KRAS mutations and other driver gene-positive subjects, they must have received at least first-line approved targeted therapy(if any) and are assessed by researchers that they hardly benefit from existing targeted therapies.
4. Has adequate organ functions, and had no blood transfusion, Erythropoietin (EPO), colony stimulating factor (CSF) or other supportive medical treatment within 14 days prior to the first dosing of GEC255.
5. Has estimated survival period ≥ 3 months.
6. Fertile female subjects must have negative serological test for pregnancy. All subjects must agree to take contraceptive measures from Informed Consent Form (ICF) signing till 3 months after last treatment.
7. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 1.

Exclusion Criteria:

1. Has received KRAS inhibitor treatment (for second part only).
2. Participated in other interventional clinical trials 4 weeks before enrollment or within 5 half-lives of the trial drug used last time (whichever is longer) .
3. Has had any anticancer treatments, including immunotherapy, chemotherapy, or radiotherapy within 4 weeks prior to the first dose of GEC255.
4. Has gastrointestinal disorder affecting absorption (eg, gastrectomy).
5. Has significant cardiovascular disease. Male subjects with corrected QT interval (QTc) ≥ 450ms, female subject with QTc ≥ 470ms
6. Has primary central nervous system (CNS) tumor;
7. Has unstable brain metastases with meningeal metastasis, spinal cord compression, symptomatic or requiring steroid/anti-epileptic medication 4 weeks before enrollment
8. HIV positive or active infection of hepatitis B virus (HBV), hepatitis C virus (HCV), syphilis, tuberculosis
9. Allergic to ingredients of GEC255; or is currently taking medicines which strongly inhibit CYP3A4.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-11-04 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients experiencing Dose limiting toxicities (DLTs) during the Maximum tolerated dose (MTD) evaluation period for study drug in monotherapy | 28 days
  characterized by type, frequency, severity (as graded by NCI CTCAE version 5.0), timing, seriousness, and relationship to study drug(Part 1)
Determine the recommended Phase II dose (RP2D) and preliminarily to develop a suitable dosing regimen | 24 months
  Measured by the number of subjects with dose limiting toxicities
Incidence of Treatment-Emergent Adverse Events | 24 months
  Characterized by type, frequency, severity (as graded by NCI-CTCAE version 5.0), timing, seriousness
Incidence of vital signs abnormalities | 24 months
  Characterized by type, frequency, severity (as graded by NCI CTCAE version5.0), and timing,seriousness
Incidence of ECG (PR interval, QRS complex, QT corrected interval prolonged, and QT interval corrected using Fridericia's formula) abnormalities | 24 months
  Characterized by type, frequency, severity (as graded by NCI CTCAE version 5.0), and timing
Incidence of laboratory abnormalities | 24 months
  Characterized by type, frequency, severity (as graded by NCI CTCAE version 5.0), and timing

SECONDARY OUTCOMES:
All study parts, Area under the plasma concentration-time curve from time zero to time t(AUC0-t) of GEC255 | Up to 24 months
  All study parts, Area under the plasma concentration-time curve from time zero to time t(AUC0-t) of GEC255
All study parts,Area under the plasma concentration-time curve from time zero to time infinity(AUC0-∞) of GEC255 | Up to 24 months
  All study parts,Area under the plasma concentration-time curve from time zero to time infinity(AUC0-∞) of GEC255
All study parts,Area under the plasma concentration-time curve over dosing interval (AUCtau) of GEC255 | Up to 24 months
  All study parts,Area under the plasma concentration-time curve over dosing interval (AUCtau) of GEC255
All study parts,Apparent plasma clearance of drug after extravascular administration(CL/F) of GEC255 | Up to 24 months
  All study parts,Apparent plasma clearance of drug after extravascular
All study parts,Terminal half-life(t½) of GEC255 | Up to 24 months
  All study parts,Terminal half-life(t½) of GEC255
All study parts,Apparent Volume of Distribution(VZ/F) of GEC255 | Up to 24 months
  All study parts,Apparent Volume of Distribution(VZ/F) of GEC255
All study parts,Maximum concentration (Cmax) of GEC255 | Up to 24 months
  All study parts,Maximum concentration (Cmax) of GEC255
All study parts,Time to maximum plasma concentration (Tmax) of GEC255 | Up to 24 months
  All study parts,Time to maximum plasma concentration (Tmax) of GEC255
Overall response rate (ORR) per RECIST v1.1, by treatment | 24 months
  Overall response rate is defined as the proportion of patients with a Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR) according to RECIST 1.1, and will be summarized along with the corresponding 95% exact binomial confidence interval (CI)
Disease Control Rate (DCR) per RECIST v1.1 | 24 months
  The disease control rate is calculated as the percentage of patients with advanced or metastatic cancer who have achieved complete response, partial response and stable disease. It will be summarized along with the corresponding 95% exact CI
Duration of Response (DOR) per RECIST v1.1 | 24 months
  Duration of response is defined as the time from the date of the first documented response (CR or PR), to the date of first documented progression, or death due any cause. Estimates will use Kaplan-Meier method, and median DOR and corresponding 95% CI will be presented
Progression-free survival (PFS) per RECIST v1.1 | 24 months
  Per RECIST 1.1, PFS is defined as the time from the date of start of treatment to the date of the first documented progression. If patient has not had an event, PFS will be censored at the date of last adequate tumor assessment
To evaluate Overall Survival (OS) following initiation of GEC255 | 24 months
  OS is defined as the time from the date of start of treatment to the date of the death
Evaluation of gene mutations profiles | 24 months
  Evaluation of gene mutations profiles including KRAS, STK11, KEAP1 etc in cell-free DNA (cfDNA) samples by Next-generation sequencing (NGS) method at various time points during treatment until disease progression

CONTACTS AND LOCATIONS:
Overall Officials: You Lu, MD, Principal Investigator — West China Hospital
Locations (1):
- China West Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No